CLINICAL TRIAL: NCT06266286
Title: The Effects of EXOPULSE Mollii Suit on Motor Functions in Children With Cerebral Palsy (EXOCEP): A Pilot Study
Brief Title: EXOPULSE Mollii Suit & Cerebral Palsy
Acronym: EXOCEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut De La Colonne Vertebrale Et Des Neurosciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-A00233-40
Record Dates: First submitted 2024-01-16; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-11

CONDITIONS: Cerebral Palsy
Keywords: Spasticity; Motor Functions; Quality of life
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: The investigators designes a randomized crossover, sham-controlled, double- blind trial to demonstrate the improvement of motor functions and cerebral palsy related symptoms following two weeks of daily sessions of "active" versus "sham" EXOPULSE Mollii suit. A two-week washout period should be enough to prevent a potential carry- over effect.
  Two weeks after the end of this phase (phase 1), a second phase of this trial, an open label phase, will be proposed for all patients to understand the effects of EXOPULSE Mollii suit and will consist of six months of active stimulation (sessions performed on a daily basis with the same parameters used for the active session in phase 1) on cerebral palsy related symptoms.
  Summary:
  * Phase 1: randomized sham controlled crossover study (active versus sham condition)
  * Phase 2: Open label study (active condition)
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator): Active stimulation sessions will last 1 hour each.
  Exopulse Mollii suits consists of a body Garments (Jacket and Pants) and a control unit. The body Garments (Jacket and Pants) is a suit with 58 embedded electrodes that can stimulate several groups of muscles, conductive wires and connectors to a detachable control unit, whose intended purpose is to transmit electric pulses from the control unit to key nerves and corresponding muscle groups throughout the body. The control unit is a battery powered electrical device which sends low intensity electric pulses through connectors to the Body Garments which in turn transmits the pulses from the connectors to key nerves and corresponding muscle groups throughout the body.
  Interventions: Device: EXOPULSE MOLLII SUIT (active)
- Sham Comparator (Sham Comparator): In the sham condition, the control unit will be programmed to start stimulating for 1 minute then it will shut off.
  Interventions: Device: EXOPULSE MOLLII SUIT (sham)

INTERVENTIONS:
Device: EXOPULSE MOLLII SUIT (active) — Exopulse Mollii suit is a new assistive device that has been developed by Exoneural Network (initially Inerventions AB), a Swedish med-tech company. Exopulse Mollii suit is a full-body garment with integrated 58 electrodes that can transcutaneously stimulate several groups of muscles.
  This stimulation is not intended to obtain a motor effect (contraction of the muscles in question), but rather to decrease the spasticity in spastic muscles by activating the antagonistic muscles via the physiological mechanism of reciprocal inhibition. The device is CE labelled and is intended to use for reducing spasticity and improving blood circulation. The outfit is very easy to put on, it can be used for one hour every day and the analgesic effects last 24 hours or more
  Arms: Active Comparator
Device: EXOPULSE MOLLII SUIT (sham) — In the sham condition, the control unit will be programmed to start stimulating for 1 minute then it will shut off
  Arms: Sham Comparator

SUMMARY:
Spasticity is a frequent and debilitating symptom in patients with cerebral palsy. It can alter the patients' balance, mobility, as well as their quality of life (QoL). The available therapeutic strategies for treating spasticity and related symptoms are usually faced with limited efficacy and numerous side effects. For these reasons, non-invasive stimulation techniques, namely transcutaneous electric nerve stimulation using EXOPULSE Mollii suit, might be of help in this context.

DETAILED DESCRIPTION:
This work will assess the effects of the EXOPULSE Mollii suit, which is an assistance device applying non-invasive transcutaneous electrostimulation. The EXOPULSE Mollii control unit is a class IIa device, CE marked, and therefore compliant with the Medical Device Directive. Its intended use includes relaxing spastic muscles, maintaining or increasing the range of movement, activating and re-educating muscles, delaying or preventing atrophy due to disuse, increasing local blood flow, and symptomatic relief and management of chronic refractory pain.

The available interventions targeting spasticity are faced with some limitations. For instance, botulinum toxin injection does not seem to improve arm and hand capacity, walking, or quality of life. The available oral agents are challenged by their potential side effects, such as sedation, drowsiness, mental confusion, fatigue, ataxia, hallucination, insomnia, nausea, dry mouth, bradycardia, hypotension, and depression, to cite a few. Therefore, developing novel therapies would help to overcome the actual limitations. Transcutaneous Electrical Nerve Stimulation (TENS) has proven some efficacy in spasticity management. However, one should note that practical difficulties could arise when using TENS at home or in clinical practice (i.e., correctly attaching electrodes). To overcome these limitations, the EXOPULSE Mollii suit has been developed by Exoneural Network, a Swedish med-tech company. It represents an innovative approach for non-invasive electro-stimulation to reduce spasticity and improve motor function.

EXOPULSE Mollii suits consist of body Garments (Jacket and Pants) and a control unit. The body Garments (Jacket and Pants) is a suit with 58 embedded electrodes that can stimulate 40 groups of muscles, conductive wires, and connectors to a detachable control unit, whose intended purpose is to transmit electric pulses from the control unit to key nerves and corresponding muscle groups throughout the body. The control unit is a battery-powered electrical device that sends low-intensity electric pulses through connectors to the Body Garments which in turn transmits the pulses from the connectors to key nerves and corresponding muscle groups throughout the body.

EXOPULSE Mollii suit consists of transcutaneously stimulating the spastic antagonist muscles with an electric current (i.e., low frequency ~20 Hz, low intensity~2 mA), aiming to reduce muscle stiffness. This treatment method's theoretical background primarily refers to the concept of reciprocal inhibition, i.e., that sensory input from a muscle may inhibit the activation of an antagonistic muscle. Thus, the application of the EXOPULSE Mollii suit aims to stimulate a muscle, e.g., the anterior tibialis muscle to reduce reflex-mediated over-activity (i.e., spasticity) of calf muscles by inducing reciprocal inhibition.

There is growing evidence now from pilot applications of EXOPULSE Mollii suit indicating beneficial effects of using this suit on activity (i.e., mobility and gross motor function) and participation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 and 12 years.
* Having a clinical diagnosis of unilateral or bilateral spastic cerebral palsy since at least one month.
* Being able to walk freely, with slight limitation or using ancillary equipment's (Gross Motor Function Classification System (GMFCS) score ≤3).
* Having a PBS score < 45.
* Being French speaker, able to understand verbal instructions, and affiliated to the national health insurance (sécurité sociale).
* Having spasticity with a score of at least 1+ on the MAS

Exclusion Criteria:

* Being included in another research protocol during the study period
* Being unable to undergo medical monitor for the study purposes due to geographical or social reasons
* Having contraindications to wearing EXOPULSE Mollii suit (i.e., implanted electronic medical devices or equipments which can be disrupted by magnets including ventriculoperitoneal shunts and intrathecal baclofen pumps, electronic life support equipment or high-frequency operation equipment, as well as well electrocardiography equipment or cardiac stimulator)
* Having a change in the pharmacological therapy over the last three months
* Suffering from other somatic or neuropsychiatric diagnoses (e.g., arrhythmias, uncontrolled epilepsy, diseases causing osteoarticular and muscular pain, skin diseases).
* Suffering from a cutaneous disease
* Using another medical device
* Being part of other protected populations as defined in articles L. 1121-5, L. 1121 6,1121-8 and L. 1122-1-2 of the Public Health Code

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in balance using the PBS (Pédiatric Balance Scale) before and after active and sham stimulation | This will be assessed at baseline (day 1), 2 weeks, 4 weeks, 6 weeks and 8 weeks
  Balance will be assessed using the 14-item PBS which has well psychometric properties in pediatric patients with cerebral palsy. The scale rates the balance using 56 points, with higher scores indicating better balance abilities.

SECONDARY OUTCOMES:
Evaluation of the cumulative effects of EXOPULSE Mollii suit on balance using the PBS | This will be assessed at 8 weeks, at 12 weeks, and at 32 weeks of using EXOPULSE Mollii suit
  Balance will be assessed using the 14-item PBS which has well psychometric properties in pediatric patients with cerebral palsy. The scale rates the balance using 56 points, with higher scores indicating better balance abilities.
Evaluation of the effects of EXOPULSE Mollii suit on spasticity using the Modified Ashworth Scale (MAS) | This will be assessed at Day 1, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 12 weeks, and at 32 weeks of using EXOPULSE Mollii suit
  It will be evaluated by examiners using the Modified Ashworth Scale (MAS; scores ranging from 0 to 4 which respectively corresponds to normal muscle tone and rigidity, which has been frequently used in clinical settings to rate muscular tone
Evaluation of the effects of EXOPULSE Mollii suit on mobility using the Timed Up and Go test (TUG) | This will be assessed at Day 1, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 12 weeks, and at 32 weeks of using EXOPULSE Mollii suit
  The score is expressed as the time (in seconds) required to perform sequential motor tasks (standing up from the chair, walking to the line on the floor at a normal pace, turning, walking back to the chair at a normal pace and finally sitting down).
Quality of life will be measured using the EuroQol 5 dimensions quality of life questionnaire for youth (EQ-5D-Y) | This will be assessed at Day 1, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 12 weeks, and at 32 weeks of using EXOPULSE Mollii suit
  This variable will be measured using the EuroQol 5 dimensions quality of life questionnaire for youth (EQ-5D-Y), a scale developed by EuroQoL group for the pediatric population and has good psychometric properties in children and adolescent. EQ-5D-Y evaluates five dimensions: anxiety/depression, mobility, pain/difficulty, selfcare, and usual activities. The score of each dimension is calculated by assigning a numerical value to each response level (i.e., 1 for "no problems", 5 for "extreme problems"/"unable to") and summing these values across the five items, resulting in a score raning from 5 (no problems on any dimension) to 25 (extreme problems on all dimensions).
Pain will be assessed using the Pain Scale Chart (PSC) | This will be assessed at Day 1, 2 weeks, 4 weeks, 6 weeks, 8 weeks,12 weeks, and at 32 weeks of using EXOPULSE Mollii suit
  Patients suffering from pain are asked to fill in the Pain Scale Chart (PSC) scored from 0 to 10 for pain. 0 meaning no pain and 10 meaning the worst pain experienced.
Evaluation of overall improvement using the Clinical Global Impression (CGI) | This will be assessed at Day 1, 2 weeks, 4 weeks, 6 weeks, 8 weeks,12 weeks, and at 32 weeks of using EXOPULSE Mollii suit
  It's consisting of 7-point scale ranging from "very much improved since the initiation of treatment" to "very much worse since the initiation of treatment" (from 1 to 7)

CONTACTS AND LOCATIONS:
Overall Officials: Samar S AYACHE, MD, PhD, Study Director — Clinical Neurophysiology department, Henri Mondor Hospital, Creteil, France
Locations (4):
- France (4):
  - Centre Hospitalier Intercommunal D'Aix Pertuis, Aix-en-Provence
  - Centre Medico Chirurgical de Readaptation Des Massues, Lyon
  - Centre de Sante Rossetti, Nice
  - Centre de Readaptation Pediatrique D'Oleron, Saint-Trojan-les-Bains

IPD SHARING:
Plan to Share IPD: No